CLINICAL TRIAL: NCT07037810
Title: A Randomized Non-inferiority Trial to Compare Multiple Daily Injections With Carbohydrate Counting or With Simplified Qualitative Meal-Size Estimation in Type 1 Diabetes: A Randomized Controlled Crossover Design.
Brief Title: Compare Multiple Daily Injections With Carbohydrate Counting or With Simplified Qualitative Meal-Size Estimation in Type 1 Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RA HM-2024-14
Record Dates: First submitted 2025-06-04; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 diabetes; carbohydrate counting; clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Placebo Comparator): MDI+FreeStyle Libre 2+ Carb counting
  Interventions: Other: Carb counting
- Experimental (Experimental): MDI+ FreeStyle Libre 2 +iBolus
  Interventions: Device: iBolus

INTERVENTIONS:
Device: iBolus — MDI+ FreeStyle Libre 2 +iBolus
  Arms: Experimental
Other: Carb counting — MDI+FreeStyle Libre 2+ Carbcounting
  Arms: Usual care

SUMMARY:
Type 1 diabetes (T1D) is an autoimmune disease characterized by loss of Beta cells in the pancreas, thus exogenous insulin is the mainstay of the management of it. Currently insulin is taken either in fixed doses for meals or variable doses via carbohydrate counting method. Fixed insulin dosing regimen may result in hyperglycemia or hypoglycemia if the insulin dose was mismatched with the ingested meal. Carbohydrate counting method was found to be superior to the fixed dosing insulin regimen. However, literature search revealed that there is a tendency to underestimate the amount of carbohydrates in meals when carbohydrate counting method was used.

To assist people with diabetes in making better decisions regarding their diabetes care, new technological tools were introduced. Among those tools a novel learning algorithm (LA) that was created to assist in optimizing carbohydrate ratio for patients with T1D on multiple daily injection (MDI) therapy.

Therefore, in this study we aim to investigate the non-inferiority of simplified qualitative meal size estimation for insulin dosing compared to carbohydrate counting method through a mobile application that is designed with the purpose of alleviating the burden of carbohydrate counting for people with T1D on multiple daily injection regimen in a randomized controlled trial with cross-over design.

Sub-Study:

Due to the significant changes in participants' diets during the month of Ramadan, none of the two interventions will be conducted during the month of Ramadan (i.e., no intervention will start in the three months preceding the month of Ramadan). However, those participants who wish to fast may enroll in an exploratory sub-study during the month of Ramadan. The sub-study will be a two-arm, crossover study in which each participant will undergo two weeks of conventional therapy and two weeks of using the McGill iBolus mobile application to adjust their basal dose and carbohydrate ratio. The primary hypothesis of this exploratory sub-study that the McGill iBolus mobile application will improve glucose control, as measured by the percentage of time spent in target range (3.9-10 mmol/L), in patients with type 1 diabetes who fast during the month of Ramadan. Note that participants may opt to participate in this sub-study and not the main study, in which case they will not be counted towards the recruitment goal of the main study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 21 years of age.
2. Clinical diagnosis of T1D for at least 12 months. The diagnosis of T1D is based on the investigator's judgment; C-peptide level and antibody determinations are not needed.
3. On MDI therapy.
4. Previously trained to count carbohydrates through a structured education program or known to perform carbohydrate counting by their educator/ dietitian.
5. Baseline HbA1c value ≥ 7.5% and < 11% (up to 7 days before or after screening)

Exclusion Criteria:

1. Serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
2. Failure to comply with the study protocol or with team's recommendations.
3. Injection of isophane insulin (NPH) or any intermediate-acting insulin.
4. More than 1 slow-acting injection and unwilling to switch to once a day for the study
5. Current or ≤ 1 month use of other antihyperglycemic agents (SGLT2, GLP-1, Metformin, Acarbose, etc.).
6. Pregnancy.
7. Severe hypoglycemic episode within one month of admission.
8. Severe diabetic ketoacidosis episode within one month of admission.
9. Clinically significant nephropathy, neuropathy, or retinopathy as judged by the investigator.
10. Conditions that may interfere with accurate HbA1c levels: clinically significant anemia, hemoglobinopathy, or a recent blood transfusion as judged by the investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 12 month
  Time spent in glucose target range 3.9-10 mmol/L (70-180 mg/dl)

SECONDARY OUTCOMES:
Secondary endpoint | 12 month
  Time spent in glucose range will be measured in percentage. Between 3.9 and 7.8 mmol/L; below 3.9 mmol/L; below 3.3 mmol/L; below 2.8 mmol/L; above 7.8 mmol/L; above 10 mmol/L; above 13.9 mmol/L; above 16.7 mmol/L.
Secondary endpoint | 12 month
  HbA1c (%)
Secondary endpoint | 12 month
  Percentage of overnight time (23:00-7:00) of sensor glucose levels. Between 3.9 and 7.8 mmol/L; below 3.9 mmol/L; below 3.3 mmol/L; below 2.8 mmol/L; above 7.8 mmol/L; above 10 mmol/L; above 13.9 mmol/L; above 16.7 mmol/L.
Secondary endpoint | 12 month
  Percentage of daytime (7:00-23:00) of sensor glucose levels. Between 3.9 and 7.8 mmol/L; below 3.9 mmol/L; below 3.3 mmol/L; below 2.8 mmol/L; above 7.8 mmol/L; above 10 mmol/L; above 13.9 mmol/L; above 16.7 mmol/L.
Secondary endpoint | 12 month
  Standard deviation of glucose levels as a measure of glucose variability
Secondary endpoint | 12 month
  Total insulin delivery (Unit/day)
Secondary endpoint | 12 month
  Mean sensor glucose level during, the overall study period, daytime period, overnight period

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa Al Ozairi, MD, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No